CLINICAL TRIAL: NCT02888951
Title: Do Standard Preoperative Fasting Instructions Ensure an Empty Stomach in Diabetic Patients? A Prospective Comparative Cohort Study
Brief Title: Gastric Ultrasound of Diabetic and Non-Diabetic Patients Following Preoperative Fasting Instructions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 15-8808-AE
Record Dates: First submitted 2016-08-22; First posted 2016-09-05 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2019-02

CONDITIONS: Diabetes; Diabetes Mellitus; Diabetes Mellitus Type 1; Diabetes Mellitus Type 2
Keywords: Diabetes; Diabetes Mellitus; Gastric Ultrasound; Preoperative fasting; Empty Stomach; Gastric Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic Group: A group of diabetic patients who have fasted for at least 8 hours undergoing an elective surgical procedure.
- Non-Diabetic Group: A group of non-diabetic patients who have fasted for at least 8 hours undergoing an elective surgical procedure.

SUMMARY:
This study evaluates the amount of fluid remaining in the stomach of diabetic patients after a standard fasting period, and compare it with non-diabetic patients coming for elective surgical procedures.

DETAILED DESCRIPTION:
Any surgical procedure carries an inherent risk of pulmonary aspiration. Food or liquid from the stomach might be forced back up the throat from where it could enter the lungs (aspiration) resulting in serious complications prolonging the hospital stay or in extreme circumstances death.

The risk of this is slightly higher in diabetics when compared to non-diabetics as the emptying of contents from the stomach is slightly delayed. This is why people going for surgery are asked not to eat for a specific time before their surgery. Anesthesiologists have recently developed an ultrasound test to determine if there is content in a patient's stomach and how much. This test involves an ultrasound examination of the abdomen and taking some measurements on the ultrasound screen.

This study aims to evaluate the amount of fluid remaining in the stomach of diabetic patients after a standard fasting period, and compare it with non-diabetic patients coming for elective surgical procedures. The investigators also aim to find an association between the type and duration of diabetes mellitus with residual gastric volume. Episodes of intra-operative regurgitation, vomiting or aspiration will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery aged 18 to 85 years
* American Society of Anesthesia physical status classification I to III
* Body mass index < 40 kg/ cm2.

Exclusion Criteria:

* Pregnancy (currently or within the past 3 months)
* Previous surgery of the upper gastrointestinal tract
* Achalasia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be patients whom are scheduled to undergo elective surgical procedures requiring preoperative fasting period of at least 8 hours. 240 patients will be recruited in total. One cohort consisting 120 patients will be diabetic (type 1 or 2). The other cohort consisting of 120 patients will be non-diabetic.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-08; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Volume of Gastric Contents | Less than two hour prior to surgery
  A "full stomach" is defined as one containing a) solid or thick fluid content or b) > 1.5 mL/kg of clear fluid.
  There are 4 categories regarding gastric contents:
  1. Empty Stomach
  2. Grade 1 Clear Fluid (fluid only observed in supine or right lateral decubitus position)
  3. Grade 2 Clear Fluid (fluid only observed in both supine and right lateral decubitus position)
  4. Solid

SECONDARY OUTCOMES:
Distribution of baseline gastric volume in fasted diabetic and non-diabetic patients | Less than two hour prior to surgery
  Characterize the distribution of baseline gastric volume in fasted diabetic and non-diabetic patients
Define the upper limit of normal fasting gastric volume defined as the 95th percentile | Less than two hour prior to surgery
  Define the upper limit of normal fasting gastric volume defined as the 95th percentile
Duration and degree of glycemic control with baseline gastric fluid volume amongst diabetic patients | Less than two hour prior to surgery
  To study the association between type of diabetes mellitus (I or II), duration and degree of glycemic control with baseline gastric fluid volume
Gastric volume of diabetic patients in relation with the medication/therapy used manage their diabetes. | Less than two hour prior to surgery
  To study the relationship between gastric volume in diabetic patients in relation with which medication and/or treatment they use to manage their diabetes. Examples of medication or treatment include; pharmaceutical hypoglycemics, insulin, or diet controlled.
Episodes of intra-operative regurgitation, vomiting or aspiration | Intraoperative
  Episodes of intra-operative regurgitation, vomiting or aspiration

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided at this time whether data will be shared.